CLINICAL TRIAL: NCT02787447
Title: A Phase II Trial of Hypofractionated Radiotherapy Combined With Thymosin for Metastatic NSCLC Patients Who Showed Stable Disease After First Line TKI Therapy
Brief Title: Radiotherapy Combined With Thymosin for Metastatic NSCLC Patients Who Showed Stable Disease After First Line TKI Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZCH-2016-09
Record Dates: First submitted 2016-04-23; First posted 2016-06-01 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Lung Adenocarcinoma
Keywords: Hypofractionated Radiotherapy; Thymosin Alpha 1; Lung Adenocarcinoma; Tyrosine Kinase Inhibitors
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Gefitinib; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): After 3 mos TKI, patients showed stable disease take TKI, radiotherapy and thymosin alpha 1 till tumor progression.
  Interventions: Drug: TKI; Radiation: Thoracic Hypofractionated Radiotherapy; Drug: Thymosin Alpha 1

INTERVENTIONS:
Drug: TKI — Gefitinib 250mg po qd or Erlotinib 150mg po qd or Icotinib 125mg po tid
  Other Names: Gefitinib/Erlotinib/Icotinib
Radiation: Thoracic Hypofractionated Radiotherapy — 40-45 Gy/5-15f
Drug: Thymosin Alpha 1 — Initiating thymosin alpha 1 therapy(1.6mg, qd, d1-d14;1.6mg, biw, d15-d90) at the second week of radiotherapy.
  Other Names: Zadaxin

SUMMARY:
The investigators postulated that the exploitation of the pro-immunogenic effects of radiotherapy with thymosin might result in abscopal responses among patients with metastatic cancer. The research is designed to evaluate the efficacy and toxicity of patients treated with hypofractionated radiotherapy combined with thymosin alpha 1. An exploratory biomarker analysis in blood and tumor samples is also planned.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic lung adenocarcinoma harboring sensitizing EGFR mutations (L858R, exon 19 deletion), and showed stable disease after 3 months TKI, evaluated twice by PET/CT scan, brain MRI, and abdomen ultrasound (≥3 measurable lesions, and these lesions haven't received local therapy)
* Age 18 years or older
* ECOG Performance Status 0-2
* Adequate bone marrow, liver and renal function, as specified below: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L; Hemoglobin ≥ 8 g/dL; Platelets ≥ 100 x 109/L; Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) ; AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present; Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter
* Patients and their family signed the informed consents

Exclusion Criteria:

* Received chemotherapy before TKI therapy
* Brain parenchyma or leptomeningeal disease
* Concurrent malignancies other than non-melanoma skin cancer that require active ongoing treatment
* Any medical co-morbidities that would preclude radiation therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with an abscopal response assessed at 1-6 months after the radiation therapy | 1-6 months
  To assess the proportion of patients with an abscopal response (defined as at least a 30% decrease in the longest diameter of the best responding abscopal lesion) at 1-6 months after the radiation therapy

SECONDARY OUTCOMES:
To assess the short-term quality of life (QOL) | 4 months
  FACT-E score at the 4 months after docetaxel consolidation therapy
Rate of CTCAE grade 2 or higher radiation pneumonitis | 1 years
  The investigators will assess the rate of symptomatic radiation pneumonitis in patients who received the radiation therapy
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China